CLINICAL TRIAL: NCT06074952
Title: Comparing the Color Stability of Acrylic Denture Teeth in Different Staining Solutions-In Vitro Experimental Trial
Brief Title: Comparing the Color Stability of Acrylic Denture Teeth in Different Staining Solutions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Huda Adil, Principal investigator, Altamash Institute of Dental Medicine
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: AltamashHC
Record Dates: First submitted 2023-09-11; First posted 2023-10-10 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Color Stability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A- Control group (Other): Control group will use distilled water as a control medium
  Interventions: Other: Aquafina(water), Coca-cola(coke), Tapal(tea), Shan(turmeric), Krikland(honey)
- Group B- Study group (Other): In this group, 4 sub-groups will be made in which acrylic teeth of Welbite brand will be immersed in tea, coke, turmeric, and honey solutions.
  Interventions: Other: Aquafina(water), Coca-cola(coke), Tapal(tea), Shan(turmeric), Krikland(honey)
- Group C- Study group (Other): In this group, 4 sub-groups will be made in which acrylic teeth of the Huge Kaili brand will be immersed in tea, coke, turmeric, and honey solutions.
  Interventions: Other: Aquafina(water), Coca-cola(coke), Tapal(tea), Shan(turmeric), Krikland(honey)

INTERVENTIONS:
Other: Aquafina(water), Coca-cola(coke), Tapal(tea), Shan(turmeric), Krikland(honey) — Distilled water will be used as a control medium in the control group. In group B, tea, coke, turmeric, and honey solutions will be used. In group C, tea, coke, turmeric, and honey solutions will be used.

SUMMARY:
The purpose of this (In Vitro Experimental Trial) is to assess (the color stability of acrylic denture teeth) in( different staining solutions) at (time intervals).

The (acrylic denture) teeth will be immersed in (staining solutions) and the values will be recorded at (different time intervals).

Three groups will be made:

* Group A- Control group
* Group B- Study group
* Group C- Study group

DETAILED DESCRIPTION:
In this study, two brands of acrylic denture teeth will be used for comparing the color stability in different staining solutions at time intervals. Identified staining substances which are tea, coke, and turmeric will be used for the staining effect evaluation. Honey solution will be used for the first time as a staining agent because honey consumption is most common in all the age groups due to its therapeutic effects. In this study, all the color values will be measured by using Portable Colorimeter (NH300, China).These values will be measured before the immersion and then after 7-days, 15-days and 21-days interval after the immersion in the solutions.

The purpose of this study is to assess the color stability of acrylic denture teeth in different staining solutions at time intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Maxillary central incisor teeth
2. Teeth with normal flat labial surfaces
3. Inter-penetrating polymer network (IPN) teeth

Exclusion Criteria:

1. Posterior teeth
2. Teeth with stains
3. Fractured and worn-out teeth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Color stability | The acrylic teeth will be measured at 7-days, 15-days, and lastly at 21-days interval.
  Color stability of acrylic denture teeth in different staining solutions will be measured by using colorimeter at different time intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Naseer Ahmed, BDS,FCPS, Study Director — Altamash Institute of Dental Medicine
Locations (1):
- Altamash Institute of Dental medicine and Karachi University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No